CLINICAL TRIAL: NCT02589249
Title: The Effect of AyuFlex® Dietary Supplementation on Joint Mobility, Comfort and Functional Capacity in Healthy Overweight Subjects
Brief Title: The Effect of AyuFlex® Supplementation on Joint Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Applied Health Sciences, LLC (Industry)
Collaborators: Natreon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NATAF-001-2015
Record Dates: First submitted 2015-10-26; First posted 2015-10-28 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Arthralgia
MeSH Terms: conditions — Arthralgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): placebo
  Interventions: Dietary Supplement: Placebo
- AyuFlex1 (Active Comparator): AyuFlex1 (500 mg/d)
  Interventions: Dietary Supplement: AyuFlex
- AyuFlex2 (Active Comparator): AyuFlex2 (1000 mg/d)
  Interventions: Dietary Supplement: AyuFlex

INTERVENTIONS:
Dietary Supplement: AyuFlex — Active product
  Arms: AyuFlex1; AyuFlex2
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this 12-week, prospective study is to determine the effects of oral supplementation with AyuFlex® (an over-the-counter dietary supplement) on joint mobility, joint comfort and functional capacity in healthy overweight subjects.

DETAILED DESCRIPTION:
This interventional study is a 12-week, randomized, double-blind, placebo and dose-response controlled clinical trial (in 3 parallel groups) of male and female subjects without active osteoarthritis of the knee to be recruited at a single investigational center in the U.S. A two-week placebo lead-in period will precede the study to enhance statistical power. One-hundred and five (105) overweight, apparently healthy subjects, pre-screened using health history questionnaires, vital signs, blood work and a standardized lower extremity exercise performance test will be randomized to one of three groups for 84 days: placebo, AyuFlex1 (500 mg/d) or AyuFlex2 (1000 mg/d). AyuFlex is an organic, non-GMO, over-the-counter joint health product derived from the edible fruits of Terminalia chebula.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers >35 to <70 years of age.
* Non-smoker.
* Body Mass Index (BMI) greater than 30 kg/m2 and less than 45 kg/m2 at screening.
* Willing to maintain current background dietary and physical activity pattern throughout study period.
* Knee joint:

  * No knee joint discomfort at rest.
  * Experience knee joint discomfort with activity or exercise within the last 2 weeks of at least 30 mm out of 100mm on VAS rating for "knee discomfort with activity or exercise at any time over the last 3 weeks".
  * Must achieve a rating of at least 30mm on a 100mm VAS at any point throughout the standardized lower extremity exercise performance screening test (Screening test = 3 sets of 10-12 repetitions on seated knee extension machine + 3-minute walk test at maximal walking velocity).
* Non-pregnant, non-lactating females who agree to use effective contraceptive methods throughout the course of the study.
* Females of childbearing potential must agree to use one of the following acceptable birth control methods:

  1. Surgically sterile (hysterectomy or bilateral oophorectomy);
  2. Surgically sterile (bilateral tubal ligation with surgery at least 6 weeks prior to study initiation);
  3. Intrauterine device (IUD) in place for at least 3 months;
  4. Abstinence (not having sexual intercourse);
  5. Barrier method (condom or diaphragm) with spermicide for at least 14 days prior to screening and through study completion;
  6. Vasectomized partner.
* Able to understand study procedures and provide signed informed consent, and authorizes release of relevant health information to study investigator.
* Normally active and otherwise judged to be in good health on the basis of medical history and physical examination.
* Females of childbearing potential must have a negative urine pregnancy test at screening.

Exclusion Criteria:

* Subjects with an established diagnosis of inflammatory joint disorder or osteoarthritis per ACR (American College of Rheumatology) guidelines.
* Currently taking, or chronic use within 30 days of anti-inflammatory supplements, Boswellia, Curcumin, Omega-3 fatty acids, Glucosamine, Chondroitin, MSM, or Collagen supplements of any type.
* Daily use of NSAIDs (non-steroidal anti-inflammatory drugs); however, daily use of 81 mg of aspirin (not > 81 mg) for cardioprotection is allowed.
* Upon physical screening by the medical staff, any subject with signs of overt nutrient deficiencies or metabolic abnormalities such as anemia. This will also need to be included in the screening assessment.
* Subjects with a history of knee or hip joint replacement surgery, or any hip or back pain which interferes with walking or exercise testing utilized throughout the study.
* Glucocorticoid (Corticosteroid) injection, hyaluronic acid injection, prolotherapy, or PRP (platelet rich plasma) injection, bone marrow or other regenerative injection in affected knee within 6 months prior to enrollment in study.
* Individual has any recent illness or condition (within 6 months of screening) that the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, or might confound the interpretation of the study results or put the person at undue risk.
* Known or suspected pregnancy, planned pregnancy, or lactation.
* If the subjects has been treated for any psychiatric illness or hospitalized for such within the past year, upon PI discretion, will be excluded from the study.
* History of allergic reaction or known sensitivity to Terminalia chebula or other chemically related botanical/ herbal products or supplements.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the Investigator, could contraindicate the subject's participation in this study.
* Vital sign abnormalities (seated, resting systolic blood pressure lower than 90 or higher than 150 mmHg, diastolic blood pressure lower than 50 or higher than 100 mmHg, or heart rate less than 50 or more than 110 bpm) at screening.
* History or clinically significant gastrointestinal disorder, (eg, inflammatory bowel diseases), presence of any gastrointestinal pathology, persistent gastrointestinal symptoms (eg, diarrhea, vomiting), liver or kidney disease, gastric bypass, gastric stapling, use of Lapband, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of dietary supplements.
* History of active neurological, endocrine, cardiovascular, pulmonary, hematological, immunologic/ autoimmune, psychiatric, or metabolic disease that is considered clinically significant by the PI.
* Recent history of (within past 12 months), or strong potential for, alcohol or substance abuse. Alcohol abuse will be defined as >14 drinks per week (1 drink = 12 oz beer, 5.0 oz wine, or 1.5 oz distilled spirits).
* Exposure to any investigational agent or drug product within 30 days prior to study entry.
* Subjects who have any physical disability which could interfere with their ability to perform the functional performance measures included in this protocol.
* Individual has a condition the Investigator believes would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results or put the patient at undue risk.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-11; Primary Completion 2017-02-07 (Actual); Study Completion 2017-02-07 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Change in score from Day 0 to day 14, 42, and 84
Visual Analogue Scale scores for discomfort, mobility, disability | Change in score from Day 0 to day 14, 42, and 84

SECONDARY OUTCOMES:
Inflammatory biomarkers | Change from Day 0 to 84
  tumor necrosis factor-alpha, c-reactive protein, and cartilage oligomeric matrix protein
6 minute walk test | Change in score from Day 0 to day 14, 42, and 84
  Total distance covered in 6 minutes
Range of motion of pain-free knee flexion/extension | Change from Day 0 to 84
Blood chemistry | Change from Day 0 to 84
  Comprehensive metabolic panel, CBC, lipid panel
Vital signs | Change in score from Day 0 to day 14, 42, and 84
  Resting heart rate and blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Tim N Ziegenfuss, PhD, Principal Investigator — The Center for Applied Health Sciences

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lopez HL, Habowski SM, Sandrock JE, Raub B, Kedia A, Bruno EJ, Ziegenfuss TN. Effects of dietary supplementation with a standardized aqueous extract of Terminalia chebula fruit (AyuFlex(R)) on joint mobility, comfort, and functional capacity in healthy overweight subjects: a randomized placebo-controlled clinical trial. BMC Complement Altern Med. 2017 Oct 2;17(1):475. doi: 10.1186/s12906-017-1977-8. PMID 28969626